CLINICAL TRIAL: NCT07154004
Title: Clinical Study on Epidermal Cell Renewal Efficacy of 5 Products
Brief Title: The Sponsor Assigns Test Products to Six Skin Areas According to a Concealed Randomization Schedule; Neither the Evaluating Physicians Nor the Participants Know Which Product is Applied to Which Site, Preventing Bias.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BEIJING YUANBEN INFORMATION CONSULTING CO., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UB24CL09012
Record Dates: First submitted 2025-08-21; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: No Protrusion; No Open Wound; No Severe Allergic Reaction; No Scar; No Tattoo; No Significant Skin Defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental)
  Interventions: Other: Test Serum 897222 210; Other: Test Serum 897222 212; Other: Test Serum 897250 39; Other: Test Serum 897250 102D; Other: Test Serum 774569 67

INTERVENTIONS:
Other: Test Serum 897222 210 — Repeated application
Other: Test Serum 897222 212 — Repeated application
Other: Test Serum 897250 39 — Repeated application
Other: Test Serum 897250 102D — Repeated application
Other: Test Serum 774569 67 — Repeated application

SUMMARY:
This is a single-center, double-blind, randomized, and controlled study. The sponsor keeps the allocation of products to the six test sites confidential. Neither the evaluating physicians nor the participants know which product is applied to which site.

The investigator will recruit 33 Chinese female participants and aim to complete the study with at least 30 of them. Each participant will be followed for 23 consecutive days.

* **Day 0**: After signing informed consent and passing screening, a staff member performs a dansyl chloride patch test. The reagent is placed in a Finn chamber, applied to the inner forearm, and sealed with waterproof tape.
* **Day 1 (≥20 h later)**: Participants return to the site. The patches are removed, photographs are taken, and the designated test products are applied to the marked areas.
* **Days 2-21**: Participants visit daily for product application by staff. After each use they report any adverse reactions, specifying symptoms, severity, location, and duration. Starting on Day 1, a dermatologist performs daily clinical scoring and photography of the test areas.

Throughout the study, participants must avoid sunscreen and any other skin-care products on the inner forearms. From Day 0 to Day 1 they may not bathe or wet the forearms; during the remaining application period they may shower but must not rub or scrub the inner forearms, and must still refrain from any other topical products.

ELIGIBILITY:
Inclusion Criteria:

- 1) Chinese physically healthy female participants, aged between 18 and 65 years old; 2) All skin types (including dry, normal, oily, and combination); 3) Have no significant skin defects, scars, tattoos, protrusions, open wounds, or other factors that would affect the evaluation on the inner side of the forearm skin; 4) Have no severe allergic reactions to the testing reagents containing dansyl chloride; 5) Agree to avoid swimming, prolonged sun exposure, sauna, and steam baths during the study period; 6) Agree to discontinue the use of any other cleansing and skincare products on the forearm during the study period; 7) Willingness to read, write and sign an informed consent form to demonstrate willingness and ability to participate; 8) Willingness to comply with all requirements of the research protocol; 9) Have no reason assessed by the investigators as unsuitable for participation in the testing; 10) Intends to complete the study and is willing and able to follow all study instructions.

11) Subjects who could comply with standards during the whole study that refrain from the use of towel, bath ball or any other bath sponges on the forearm.

Exclusion Criteria:

* 1) Undergoing dermatological treatment or those who have taken whitening or anti-aging dietary supplements within the past month; 2) Have allergies to skincare products, soap, alcohol, fragrances, or medications; 3) Have used antihistamines within the past week or immunosuppressants within the past month; 4) Have applied any anti-inflammatory drugs to the test area within the past two months; 5) Have skin conditions such as psoriasis, eczema, dermatitis, skin cancer, etc.; 6) Insulin-dependent diabetes patients; 7) Undergoing treatment for asthma or other chronic respiratory diseases; 8) Have received cancer chemotherapy within the past 6 months; 9) With immunodeficiency or autoimmune diseases; 10) Breastfeeding or pregnant women; 11) Have undergone bilateral mastectomy and bilateral axillary lymph node dissection; 12) With facial erythema, follicular papules, sunspots, wounds, abrasions, tattoos, acne, or any other conditions that may affect the evaluation of test results; 13) With high sensitivity; 14) Have participated in intense outdoor activities or travel that may cause skin damage due to sun exposure within the month prior to the test; 15) Concurrently participating in another clinical trial or who have participated in a facial clinical trial within the past three months; 16) Have applied vitamin A analogues, alpha-hydroxy acids, salicylic acid, hydroquinone, or prescription drugs (antibiotics, vitamin A analogues, alpha-hydroxy acids, and corticosteroids) within the past six months, or oral contraceptives (continuation is allowed if the same contraceptive has been used consistently for the past six months); 17) PI or experts who believe that there are other medical reasons that may affect the test results.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-21 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Clinical Grading by Dermatologist | Day 1 to Day 22
  A dermatologist should use a UV lamp to illuminate the inner side of the forearm and evaluate the fluorescence area in the target region daily from Day 1 to Day 22

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Yuanben Information Consulting Co., Ltd, Beijing, China

IPD SHARING:
Plan to Share IPD: No